CLINICAL TRIAL: NCT06401642
Title: A Study to Assess Effectiveness and Tolerability of Zavegepant as an Acute Migraine Treatment Among Those Using CGRP Targeting Preventive Medications.
Brief Title: Effectiveness and Tolerability of Zavegepant for Acute Migraine Treatment Among Those Using CGRP Targeting Preventive Medications
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Todd J. Schwedt, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-011210
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zavegepant Treatment (Experimental): Participants will receive zavegepant to treat up to 8 migraine attacks over 24 weeks.
  Interventions: Drug: Zavegepant

INTERVENTIONS:
Drug: Zavegepant — 10 mg intranasal

SUMMARY:
Zavegepant (Zavzpret) is approved for the acute treatment of migraine with or without aura in the US. The purpose of this study is to investigate the effectiveness and tolerability of zavegepant for the acute treatment of migraine attacks amongst participants who are using calcitonin gene-related peptide (CGRP) migraine preventive treatments.

DETAILED DESCRIPTION:
This is a phase IV, open-label, prospective, longitudinal clinical trial of intranasal zavegepant 10 mg, a CGRP receptor antagonist, for the acute treatment of migraine attacks amongst individuals who are concomitantly taking stable doses of CGRP targeting migraine preventive treatment (atogepant, eptinezumab, erenumab, fremanezumab, galcanezumab, rimegepant). The effectiveness and tolerability of zavegepant will be assessed in this specific participant population. Participants who are not already taking a CGRP-targeting migraine preventive treatment but who meet criteria for migraine prevention according to their clinician's discretion, will have the option to start rimegepant 75 mg every other day (qod) for two months. After two months, continued eligibility for participation in the clinical trial of zavegepant will be assessed. Those receiving rimegepant for migraine prevention through their participation in this study will have the option to receive rimegepant for up to 32 consecutive weeks.

ELIGIBILITY:
Inclusion Criteria

* Meets International Classification of Headache Disorders 3 (ICHD-3) diagnostic criteria for migraine with or without aura
* At least 18 years of age
* 2- 8 migraine attacks per month
* Participants should be on a calcitonin gene-related peptide (CGRP)-targeting preventive migraine medication on a stable dose for a) ≥2 months prior to zavegepant treatment if an oral gepant or a monoclonal antibody (mAb) injected monthly, or b) at least two treatments if a mAb injected each 3 months.

  * Atogepant
  * Eptinezumab
  * Erenumab
  * Fremanezumab
  * Galcanezumab
  * Rimegepant

Exclusion Criteria

* Primary headache disorders other than migraine (tension-type headache days are allowed)
* History of hypersensitivity reaction to zavegepant or to any of the components of zavegepant

Eligibility Notes

* Participants may have either episodic or chronic migraine.
* Prior use of zavegepant and other gepants is permitted.
* Participants can be using migraine preventive medications/treatments in addition to the CGRP-targeting preventive treatment, as long as those treatments have been stable for at least two months at the time of enrollment.

Additional Eligibility Criteria for Participants to Start on Rimegepant for Migraine Prevention

Inclusion Criteria:

• Must have 4 or more migraine days per month, on average, during the 2 months prior to the Screening Visit, according to participant self-report.

Exclusion Criteria

• History of hypersensitivity reaction to rimegepant or to any of the components of rimegepant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Headache relief in 2 hours | 2 hours
  Percentage of participants who have meaningful headache relief within 2 hours of administering zavegepant
Headache relief in 4 hours | 4 hours
  Percentage of participants who have meaningful headache relief within 4 hours of administering zavegepant
Functional disability level in 2 hours | 2 hours
  Percentage of participants with functional disability level of normal or mildly impaired within 2 hours of administering zavegepant.
Functional disability level in 4 hours | 4 hours
  Percentage of participants with functional disability level of normal or mildly impaired within 4 hours of administering zavegepant.

SECONDARY OUTCOMES:
Adverse events | Approximately 24-32 weeks
  Percentage of participants and treated migraine attacks with treatment emergent adverse events
Serious adverse events | Approximately 24-32 weeks
  Percentage of participants and treated migraine attacks with serious treatment emergent adverse events
Discontinuation due to adverse events | Approximately 24-32 weeks
  Percentage of participants who discontinue zavegepant due to adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schwedt, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Zavegepant to Treat Migraine Attacks — https://www.mayo.edu/research/clinical-trials/cls-20567120